CLINICAL TRIAL: NCT01696123
Title: Efficacy and Tolerability of MLC601 in Patients With Mild to Moderate Alzheimer Disease Who Were Unable to Tolerate or Failed to Benefit From Treatment With Rivastigmine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Amini Harandi, Dr, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBMU-1391
Record Dates: First submitted 2012-09-21; First posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Cholinesterase inhibitors; MLC601; NeuroAiD; neuroprotection; neuroregeneration
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuroaid

ARMS (1):
- MLC601 (Experimental): MLC601 (NeuroAid, Moleac Pte. Ltd, Singapore) (0.4 g per capsule) was prescribed as one capsule three times daily without an escalation dose.
  Interventions: Drug: MLC601

INTERVENTIONS:
Drug: MLC601 — It was described
  Other Names: NeuroAid

SUMMARY:
Current therapeutic approaches for the treatment of neurodegenerative diseases like Alzheimer disease (AD) offer limited and often transient symptomatic benefits to patients but do not mitigate the insidious loss of neuronal cells. In this trial the investigators will evaluate Efficacy and Tolerability of MLC601 as a neuroprotective in Patients with Mild to Moderate Alzheimer Disease who Were Unable to Tolerate or Failed to Benefit from Treatment with Rivastigmine.

DETAILED DESCRIPTION:
An 18-month open-label pilot study would be conducted at three university referral centres in Tehran, Iran. All patients are at least 50 years old, met the criteria for AD according to the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), and failed treatment with the cholinesterase inhibitor Rivastigmine for any reason. A baseline medical history will be taken and physical examination will be performed for all participants, and any comorbidities and concomitant therapies would be noted. Patients with controlled concomitant diseases, such as hypertension and diabetes, will be allowed to enter the study. Mini-Mental State Examination (MMSE)10 and Alzheimer disease assessment scale-cognitive sub scale11 (ADAS-cog) will be used to measure treatment efficacy. MLC601 will be prescribed as one capsule three times daily without an escalation dose. Safety and tolerability evaluations included physical examinations, electrocardiography, vital sign monitoring and laboratory testing weekly for the first 8 weeks and every 4 weeks thereafter. The MMSE and ADAS-cog will be recorded at each efficacy follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* at least 50 years old
* met the criteria for AD according to the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* failed treatment with the cholinesterase inhibitor Rivastigmine for any reason

Exclusion Criteria:

* uncontrolled diabetes mellitus
* hypertension
* unstable cardiac disease
* severe obstructive pulmonary disease
* renal or hepatic failure
* and/or other life threatening conditions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
changes in the Mini-Mental State Examination (MMSE) relative to baseline measurements | every 4 weeks up to 18 months
  change in the Mini-Mental State Examination (MMSE) relative to baseline measurements will be evaluated every 4 weeks up to 18 months.
changes in the cognitive subscale of the AD Assessment Scale (ADAS-cog) relative to baseline measurements | every 4 weeks up to 18 months
  change in the cognitive subscale of the AD Assessment Scale (ADAS-cog) relative to baseline measurements will be evaluated every 4 weeks up to 18 months.

SECONDARY OUTCOMES:
to measure included adverse events (AEs) | every 4 weeks
  Safety and tolerability evaluations included physical examinations, electrocardiography, vital sign monitoring and laboratory testing weekly for the first 8 weeks and every 4 weeks thereafter. AEs were defined as any sign, symptom, syndrome or disease that occurred for the first time or worsened after baseline, whether they were considered treatment related.
measuring withdrawal rate | every 4 weeks
  measuring any withdrawal rate among intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Ali Amini, M.D, Principal Investigator — Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- Loghman Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Pakdaman H, Amini Harandi A, Gharagozli K, Siavoshi F, Shirzadeh Barough S, Sharifipour E, Esfandani A, Ilkhani S, Tabatabaei FS, Sobhanian SA. A Long-term Study of NeuroAid (MLC601, MLC901) in Patients with Alzheimer's Disease; An Extension 8-year Follow-up Study. Curr Aging Sci. 2023;16(3):234-239. doi: 10.2174/1874609816666230224111759. PMID 36843256